CLINICAL TRIAL: NCT00578071
Title: A Phase I/II Study of Panitumumab, Capecitabine and Oxaliplatin Chemotherapy With External Beam Radiation Therapy for the Treatment of Resectable, Locally Advanced/Unresectable or Metastatic Esophageal Cancer
Brief Title: Phase I/II Study of Panitumumab, Capecitabine and Oxaliplatin w EBRT for Esophageal Cancer
Acronym: POXX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brian Czito (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Brian Czito, Associate Professor, Radiation Oncology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002207; SPS 151596
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-05

CONDITIONS: Cancer of the Esophagus
Keywords: esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Panitumumab; Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): panitumumab, oxaliplatin, capecitabine and EBRT
  Interventions: Drug: Panitumumab; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Drug: Panitumumab — Dose per cohort level (3.6, 4.8 or 6.0 mg/kg ), given intravenously (IV) days 1, 15 and 29 of radiation.
Drug: Capecitabine — Dose per cohort level (500, 625 or 825 mg/m2) taken by mouth twice each day of radiation
  Other Names: Xeloda
Drug: Oxaliplatin — Dose per cohort level (30, 40, or 50 mg/m2). Given IV one day each week during radiation
Radiation: Radiation Therapy (RT) — Daily for 6 weeks

SUMMARY:
The primary purpose of this trial is to define the maximum tolerated and/or recommended phase II dose of the combination of panitumumab, oxaliplatin and capecitabine in patients undergoing radiation therapy for carcinoma of the thoracic esophagus or gastroesophageal junction. An additional primary objective is to describe the frequency and nature of grade III/IV and grade I/II toxicities associated with this regimen. Secondary objectives include describing 1-year disease-free survival and overall survival rates as well as to estimate clinical and pathologic complete response rates associated with this regimen.

DETAILED DESCRIPTION:
This study has a phase I/II design. For this study the administration of panitumumab is considered investigational.

Pretreatment: Part of regular cancer care and disease staging includes Chest/Abdomen CT Scan, upper endoscopic ultrasound, PET scan, J-Tube Placement (if clinically indicated), bronchoscopy (per clinician judgment), ECG, and baseline laboratory studies.

During Treatment Weeks 1-5.5 of Radiation Therapy(RT)/Chemotherapy:

* RT (180 cGy/fx, Mon-Fri) days 1-5, 8-12, 15-19, 22-26, 29-33 and 36-38.
* Panitumumab (per dose level) days 1, 15, 29.
* Oxaliplatin (per dose level) days 1, 8, 15, 22, 29, 36.
* Capecitabine (per dose level M-F) 1-5, 8-12, 15-19, 22-26, 29-33, 36-38.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Histologically or cytologically documented squamous cell carcinoma or Siewert's classification adenocarcinoma of the esophagus or proximal stomach T1-4, N0-2, M0-1, for which bimodality treatment with chemotherapy and radiation therapy is indicated.
* Measurable Disease
* ECOG Performance Status 0-1
* Laboratory values must be as follows:
* Absolute neutrophil count > or = 2,000/mm3,
* Platelets > or = 100,000/mm3,
* Hemoglobin > 9.0,
* Total bilirubin <1.5 x institutional upper normal limit,
* Serum creatinine <1.5 x institutional upper normal limit,
* AST or ALT < 3x institutional upper normal limit,
* Magnesium equal or higher than institutional lower limit,
* Creatinine clearance Estimated > 40 ml/min,
* Calcium > lower limit of normal.
* Not pregnant or lactating. Negative pregnancy test within 72 hours prior to registration (female patients of childbearing potential). Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Life expectancy must be >3 months.
* No serious or poorly controlled medical or psychological conditions that could be exacerbated by the treatment or would seriously complicate compliance with the protocol.
* Able to swallow capecitabine (whole or crushed tablet or liquid dispersed) or patients may have a G or J tube.
* No conditions that would significantly compromise intestinal absorption of the study drugs.

Exclusion Criteria:

* Tumors extending above the level of the thoracic inlet or beyond 5 cm below the gastroesophageal junction.
* Patients with radiographic or bronchoscopic evidence of esophageal perforation.
* Patients with known evidence of brain metastases, lymphangitic lung metastases, or carcinomatous meningitis.
* Dementia or significantly altered mental status
* Major surgery within 4 weeks of the start of study treatment
* Prior chemotherapy, radiation therapy, hormonal or biologic therapy within the past 6 months.
* Subjects requiring chronic use of immunosuppressive agents (e.g., methotrexate, cyclosporine, corticosteroids)
* Currently requiring medications that may interact with the metabolism or disposition of capecitabine/5-FU: dipyridamole, folinic acid, allopurinol, trimethoprim, misonidazole, metoclopramide, flucytosine or cimetidine.
* Hypersensitivity to platinum containing compounds or capecitabine or any of the excipients of this product. Prior unanticipated severe reaction to fluoropyrimidine/platinum therapy, or known sensitivity to 5-fluorouracil/platinum containing compounds.
* Serious, uncontrolled, concurrent infection(s).
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Peripheral neuropathy > grade 1
* Any of the following within 24 weeks before randomization: clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia).
* Uncontrolled gastrointestinal ulcer within 28 days of randomization
* History of interstitial pneumonitis or pulmonary fibrosis, or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest X-ray or CT-scan
* Preexisting known bleeding diathesis or coagulopathy
* Plans to continue on or use of ketoconazole, phenytoin, phenobarbital, carbamazepine, rifampin, rifabutin or St. John's Wort, 14 days prior to randomization.
* History of hypersensitivity to tetracyclines
* Subject known to be human immunodeficiency virus positive
* Subjects known to have chronic or active hepatitis B or C infection

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czito, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: Clinical Trials at Duke Comprehensive Cancer Center — http://www.cancer.duke.edu/CTrials/index.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiation: Panitumumab, oxiplatin, capecitabine, radiation therapy
Period: Overall Study
Arm/Group | Chemoradiation
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemoradiation
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.97 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Panitumumab Maximum Tolerated Dose in Milligrams (mg)
Time Frame: 60 days
Population: Per protocol and intention to treat (ITT).
Measure: Number; unit: mg
Arm/Group | Chemoradiation
Number analyzed (Participants) | 29
mg | 3.6

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Time Frame: Within 30 days of the last day of radiation
Population: All patients who received chemoradiation.
Measure: Number; unit: participants
Arm/Group | Chemoradiation
Number analyzed (Participants) | 29
participants | 2

3. Secondary Outcome: Overall Survival Rates for the Patients Studied on This Protocol.
Description: Number of patients alive one year after completing study protocol treatment.
Time Frame: One year
Measure: Number; unit: participants
Groups:
- Arm 1 Chemoradiation: Panitumumab, oxiplatin, capecitabine, radiation therapy
Arm/Group | Arm 1 Chemoradiation
Number analyzed (Participants) | 29
participants | 18

4. Secondary Outcome: Pathological Complete Response Rates Associated With This Regimen.
Description: Absence of residual viable tumor cells at the time of surgical resection of the esophagus performed 7-9 weeks following completion of chemoradiotherapy.
Time Frame: 90 days
Population: Surgery was determined according to risk factors, patient consent and resectability.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 Chemoradiation
Number analyzed (Participants) | 20
percentage of participants | 40

ADVERSE EVENTS:
Arm/Group | Chemoradiation
Serious Adverse Events (participants affected / at risk) | 9/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation (N=29)
Atrial Fibrilation (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (3)
Febrile neutropenia (Infections and infestations) | 2 (2)
Hypersensitivity reaction (Immune system disorders) | 1 (1) — Allergic reaction.
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation (N=29)
Anorexia (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dehydration (General disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 9 (9)
Edema: Limb (General disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 11 (11)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 (7)
Hiccoughs (Gastrointestinal disorders) | 3 (3)
Infection (Infections and infestations) | 7 (7)
Potassium, serum-low (Metabolism and nutrition disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 20 (20)
Neuropathy: sensory (Nervous system disorders) | 13 (13)
Pain (Nervous system disorders) | 11 (11)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 27 (27)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2)
Thrombosis, thrombus, embolism (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 16 (16)
Weight Loss (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes